CLINICAL TRIAL: NCT02441283
Title: A Follow-up Study to Assess Resistance and Durability of Response to AbbVie Direct-Acting Antiviral Agent (DAA) Therapy (ABT-493 and/or ABT-530) in Subjects Who Participated in Phase 2 or 3 Clinical Studies for the Treatment of Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Study to Assess Resistance and Durability of Response to ABT-493 and/or ABT-530
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M13-576; 2015-000452-24 (EudraCT Number)
Expanded Access: NCT03123965 (Approved for marketing)
Record Dates: First submitted 2015-04-29; First posted 2015-05-12 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-08

CONDITIONS: Hepatitis C
Keywords: Chronic hepatitis C; Hepatitis C virus; Sustained virologic response; Hepatitis C; Direct Acting Antiviral
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — glecaprevir; pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HCV-infected Participants (No Intervention): Hepatitis C virus (HCV)-infected participants who received ABT-493 and/or ABT-530 in prior Phase 2 or 3 clinical studies with these agents for the treatment of chronic HCV and were not retreated prior to entering this study. No AbbVie study drug was administered in this study.
  Interventions: Drug: ABT-493; Drug: ABT-530

INTERVENTIONS:
Drug: ABT-493 — ABT-493 was not administered in this study. This study was a follow-up for participants who received the drug in prior studies.
  Other Names: Glecaprevir
Drug: ABT-530 — ABT-530 was not administered in this study. This study was a follow-up for participants who received the drug in prior studies.
  Other Names: Pibrentasvir

SUMMARY:
This was a long-term follow-up study to evaluate the durability of sustained virologic response (SVR), persistence of direct-acting antiviral agent (DAA) resistance, and clinical outcomes for participants who received glecaprevir (ABT-493) and/or pibrentasvir (ABT-530) in prior AbbVie Phase 2 or 3 clinical studies for the treatment of chronic hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
This was a Phase 2/3, multicenter study offered to participants who received at least one dose of an ABT-493- and/or ABT-530-containing regimen at any dose level in an eligible prior AbbVie Phase 2 or 3 study for the treatment of chronic HCV and elected to enroll in this study. The participant must have completed the follow-up period of the prior eligible AbbVie study. Participants were followed for a total of approximately 3 years after their last dose of DAA in the previous HCV clinical study. The 3 years were inclusive of any post-treatment period in the prior study, as well as any gaps between the end of the prior study and enrollment in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is male or female 18 years of age or older
2. Participant has received at least one dose of an ABT-493- and/or ABT- 530 containing regimen in a prior AbbVie hepatitis C virus (HCV) Phase 2 or 3 study
3. The interval between the last dose of the AbbVie direct-acting antiviral agent (DAA) therapy from the previous clinical study and enrollment in Study M13-576 must be no longer than 2 years for subjects who have not been retreated. Participants who have been treated with a commercially available anti-HCV treatment may be enrolled greater than 2 years after the last dose of the AbbVie DAA therapy from the previous clinical study.
4. Participant must voluntarily sign and date the informed consent form approved by an Independent Review Board or Ethics Committee prior to the initiation of any study-specific procedures.
5. Participant completed the post-treatment period of an eligible prior study.

Exclusion Criteria:

1. The investigator considers the participant unsuitable for the study for any reasons (e.g., failure to comply with study procedures in the prior AbbVie clinical study).
2. Receipt of any investigational HCV antiviral treatment after receiving ABT-493 and/or ABT-530 in the prior study.
3. Participants who experienced non-virologic treatment failure due to premature discontinuation of study drug in prior study of ABT-493/ABT-530.
4. Participation in AbbVie's Study M15-942 protocol for re-treatment for virologic failure in the prior Phase 2 or 3 study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (42):
- United States (20):
  - Digestive Health Specialists of the Southeast /ID# 136725, Dothan, Alabama
  - Felizarta /ID# 141033, Bakersfield, California
  - Southern California Res. Ctr. /ID# 141799, Coronado, California
  - Research & Education, Inc. /ID# 169591, San Diego, California
  - eStudySite San Diego /ID# 141040, San Diego, California
  - eStudySite San Diego /ID# 141047, San Diego, California
  - eStudySite San Diego /ID# 141048, San Diego, California
  - Midway Immunology and Research /ID# 169477, Ft. Pierce, Florida
  - Delta Research Partners /ID# 141028, Bastrop, Louisiana
  - Louisiana Research Ctr. LLC /ID# 141024, Shreveport, Louisiana
  - Henry Ford Health System /ID# 141039, Detroit, Michigan
  - Binghamton Gastroenterology /ID# 141026, Binghamton, New York
  - Carolinas Center for Liver Dis /ID# 155390, Statesville, North Carolina
  - Northwest Gastroenterology Cli /ID# 141036, Portland, Oregon
  - Gastro One /ID# 169478, Germantown, Tennessee
  - Quality Medical Research, PLLC /ID# 141042, Nashville, Tennessee
  - TX Clinical Research Institute /ID# 141037, Arlington, Texas
  - Inquest Clinical Research /ID# 141045, Baytown, Texas
  - TX Liver Inst, Americ Res Corp /ID# 136727, San Antonio, Texas
  - Bon Secours St. Mary's Hospita /ID# 165106, Richmond, Virginia
- Australia (6):
  - St. Vincent's Hospital, Darlinghurst /ID# 155395, Darlinghurst, New South Wales
  - St. Vincents Hospital /ID# 155394, East Lismore, New South Wales
  - Westmead Hospital /ID# 155392, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital /ID# 155396, Herston, Queensland
  - Royal Adelaide Hospital /ID# 155391, Adelaide, South Australia
  - Royal Melbourne Hospital /ID# 155393, Parkville, Victoria
- Belgium (3):
  - Cliniques Universitaires Saint Luc /ID# 155397, Woluwe-Saint-Lambert, Brussels Capital
  - CHU St. Pierre /ID# 155399, Brussels
  - UZ Leuven /ID# 155398, Leuven
- Canada (2):
  - University of Calgary /ID# 155400, Calgary, Alberta
  - Toronto Liver Centre /ID# 155401, Toronto, Ontario
- Germany (3):
  - Universitätsklinikum Frankfurt /ID# 169817, Frankfurt am Main, Hesse
  - Mauss, Schmutz, Hegener, Athma /ID# 155402, Düsseldorf
  - Gastroenterologisch-Hepatologi /ID# 169820, Kiel
- Auckland City Hospital /ID# 155403, Auckland, New Zealand
- Puerto Rico (3):
  - Gastro-Hepato & Geriatric Ctr /ID# 141060, Ponce
  - Klinical Investigations Group /ID# 141059, San Juan
  - Innovative Care P.S.C. /ID# 141061, San Juan
- United Kingdom (4):
  - The Royal London Hospital /ID# 155405, London, London, City of
  - King's College Hospital NHS /ID# 155406, London
  - St. Mary's Hospital /ID# 155404, London
  - Derriford Hospital /ID# 155407, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Poordad F, Felizarta F, Yao BB, Overcash JS, Hassanein T, Agarwal K, Gane E, Shaw D, Waters M, Krishnan P, Topp A, Burroughs M, Nevens F. Durability of sustained virological response to glecaprevir/pibrentasvir and resistance development: A long-term follow-up study. Liver Int. 2022 Jun;42(6):1278-1286. doi: 10.1111/liv.15211. Epub 2022 Mar 14. PMID 35220658

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set (FAS): all participants who received ABT-493 and/or ABT-530 in a prior Phase 2/3 study and were not retreated prior to enrolling in this study.Three participants who received retreatment prior to enrollment in this study and four participants who did not receive ABT-493 and/or ABT-530 in a prior study were excluded from the FAS.
Period: Overall Study
Arm/Group | HCV-infected Participants
Started | 377
Completed | 287
Not Completed | 90
Not completed — Withdrew consent | 15
Not completed — Lost to Follow-up | 42
Not completed — Death | 1
Not completed — Other, not specified | 32

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who received ABT-493 and/or ABT-530 in a prior Phase 2 /3 study and were not retreated prior to enrolling in this study.Three participants who received retreatment prior to enrollment in this study and four participants who did not receive ABT-493 and/or ABT-540 in a prior study were excluded from the FAS.
Groups:
- HCV-infected Participants: Hepatitis C virus (HCV)-infected participants who received ABT-493 and/or ABT-530 in prior Phase 2 or 3 clinical studies with these agents for the treatment of chronic HCV and were not retreated prior to entering this study. No AbbVie study drug was administered in this study. The baseline data presented below are values at the time of the prior study start.
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172
  Male | 205
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 328
  Black or African American | 29
  Asian | 16
  American Indian or Alaska Native | 2
  Native Hawaiian or other Pacific Islander | 1
  Multi race | 1
HCV Genotype [Count of Participants; unit: Participants]
  1 | 168
  2 | 76
  3 | 106
  4 | 14
  5 | 7
  6 | 6
Baseline Cirrhosis Status [Count of Participants; unit: Participants]
  Yes | 65
  No | 312
Treatment Status Prior to Previous Study [Count of Participants; unit: Participants] — PRS= interferon (alpha, beta, or pegylated interferon) with or without ribavirin, or sofosbuvir with ribavirin with or without interferon]; NS5A= nonstructural viral protein 5A; PI= protease inhibitor
  Participants
    Naive | 265
    PRS-experienced | 83
    NS5A-experienced/PI naive | 10
    NS5A- and PI- experienced | 12
    PI-experienced/NS5A naive | 7
Baseline HIV-1/HCV coinfection status [Count of Participants; unit: Participants]
  Yes | 7
  No | 370
Baseline injection drug use status [Count of Participants; unit: Participants]
  Yes | 181
  No | 193
  Missing | 3
Baseline HCV RNA level [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2573 (0.82900)
Study Drug Regimens Received in Prior Abbvie Study [Count of Participants; unit: Participants]
  ABT-450/r + ABT-530 + RBV-12 wks | 4
  ABT-493 200 mg QD + ABT-530 40 mg QD-12 wks | 34
  ABT-493 200 mg QD + ABT-530 80 mg QD-12 wks | 1
  ABT-493 200 mg QD + ABT-530 120 mg QD-12 wks | 57
  ABT-493 200 mg QD + ABT-530 120 mg QD + RBV-12 wks | 10
  ABT-493 300 mg QD + ABT-530 120 mg QD-8 wks | 13
  ABT-493 300 mg QD + ABT-530 120 mg QD-12 wks | 20
  ABT-493 300 mg QD + ABT-530 120 mg QD-16 wks | 1
  ABT-493 300 mg QD + ABT-530 120 mg QD + RBV-12 wks | 5
  ABT-493/ABT-530 300 mg/120 mg QD- 8 wks | 74
  ABT-493/ABT-530 300 mg/120 mg QD-12 wks | 134
  ABT-493/ABT-530 300 mg/120 mg QD-16 wks | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintained a Sustained Virologic Response (SVR) Out of Those Who Achieved SVR12 in a Prior Study With an ABT-493- and/or ABT-530-containing Regimen
Description: Maintaining a sustained virologic response (SVR) is defined as having Hepatitis C virus ribonucleic acid (HCV RNA) value consistently below the lower limit of quantification (< LLOQ) from the end of treatment in the previous study throughout Study M13-576 (this study).
Time Frame: From the end of treatment in the previous study up to 3 years post-treatment
Population: Full Analysis Set (FAS):all participants who received ABT-493 and/or ABT-530 in a prior Phase 2 /3 study and were not retreated prior to enrolling in this study.Three participants who received retreatment prior to enrollment in this study and four participants who did not receive ABT-493 and/or ABT-530 in a prior study were excluded from the FAS.
Measure: Number; unit: percentage of participants
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 376
percentage of participants | 99.5

2. Primary Outcome: Percentage of Participants Who Relapsed or Had a New Hepatitis C Virus (HCV) Infection at Any Time up to the Last Follow-up in This Study Among Participants Who Achieved SVR12 in a Prior Study With an ABT-493- and/or ABT-530-containing Regimen
Description: Relapse was defined as confirmed Hepatitis C virus ribonucleic acid (HCV RNA) greater than or equal to the lower limit of quantification (≥ LLOQ) between end of treatment and up to and including the last HCV RNA measurement collected in this study for a participant with HCV RNA < LLOQ at Final Treatment Visit who completed treatment, excluding reinfection. HCV reinfection was defined as confirmed HCV RNA ≥ LLOQ after the end of treatment in a participant who had HCV RNA < LLOQ at Final Treatment Visit, along with the post-treatment detection of a different HCV genotype, subtype, or clade compared with baseline, as determined by phylogenetic analysis of the NS3 or NS5A, and/or NS5B gene sequences.
Time Frame: From the end of treatment in the previous study up to 3 years post-treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 376
percentage of participants
  Relapse overall | 0.3
  Reinfection overall | 0.3

3. Primary Outcome: Number of Participants With Persistence of Resistance-Associated Amino Acid Variants Among Those Experiencing Virologic Failure
Description: Plasma samples for HCV resistance testing were collected at study visits. The variants in nonstructural viral protein 3 (NS3) and nonstructural viral protein 5A (NS5A) at amino acid positions of interest were analyzed by next generation sequencing relative to baseline and prototypic reference sequences.
Time Frame: From Day 1 to Month 12
Population: Participants who experienced virologic failure in previous study or in the current study with available sequencing data for NS3/4A and/or NS5A
Measure: Number; unit: participants
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 1
participants
  NS3 Variants at Months 3, 6, and 12 | 1
  NS5A Variants at Months 3, 6, and 12 | 1

4. Secondary Outcome: Number of Participants With Medical Events Related to Progression of Liver Disease or Hepatitis C Virus Infection
Description: Any events (i.e., diagnoses) related to liver disease progression and/or HCV infection considered to be clinically significant by the investigator that began or worsened after Day 1 were documented until the end of the study or initiation of re-treatment for HCV (if applicable). Significant events related to liver disease progression include the development of cirrhosis, events indicative of hepatic decompensation, (including: variceal bleeding, new ascites, spontaneous bacterial peritonitis, hepatic encephalopathy, hepato-renal syndrome, hepatic hydrothorax or other evidence of hepatic decompensation considered to be significant by the investigator), change in the Child-Pugh category (e.g., change from Child-Pugh Class A to Child-Pugh Class B), the occurrence of hepatocellular carcinoma, liver transplantation and/or death.
Time Frame: After Day 1 up to 3 years post-treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 377
Participants
  Medical events related to liver disease or HCV inf | 7
  Development of cirrhosis | 0
  Liver decompensation (Variceal bleeding) | 0
  Liver decompensation (Ascites) | 0
  Liver decomp (spontaneous bacterial peritonitis) | 0
  Liver decompensation (hepatic encephalopathy) | 0
  Liver decompensation (hepatorenal syndrome) | 0
  Liver decompensation (hepatic hydrothorax) | 0
  Liver decompensation (other [PI's discretion]) | 0
  Change in Child-Pugh Score in subject w/cirrhosis | 0
  Hepatocellular carcinoma (HCC) | 5
  Liver transplantation occurred | 0
  Death | 0
  Regenerated node in the liver | 1
  Cholangiocarcinoma/differentiated adenocarcinoma | 1

5. Secondary Outcome: Mean Concentration of Interferon Gamma-induced Protein 10 (IP-10) Over Time
Description: A plasma sample for IP-10 testing was collected at study visits for all participants, until the end of the study or initiation of re-treatment for HCV (if applicable). IP-10 is used to assess liver fibrosis in participants with chronic liver disease.
Time Frame: From Day 1 up to 3 years post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 374
ng/L
  Day 1 | 146.884 (116.6272)
  Month 3: number analyzed (Participants) | 363
  Month 3 | 147.606 (118.5143)
  Month 6: number analyzed (Participants) | 336
  Month 6 | 148.959 (119.0047)
  Month 12: number analyzed (Participants) | 1
  Month 12 | 224.400
  Month 18: number analyzed (Participants) | 7
  Month 18 | 133.300 (50.2647)
  Month 24: number analyzed (Participants) | 234
  Month 24 | 140.185 (97.2769)
  Month 30: number analyzed (Participants) | 88
  Month 30 | 164.244 (276.9176)
  Month 36: number analyzed (Participants) | 1
  Month 36 | 120.600

6. Secondary Outcome: Mean FibroTest Score Over Time
Description: A serum sample for FibroTest evaluation was collected at study visits for all participants, until the end of the study or initiation of re-treatment for HCV (if applicable). FibroTest uses six biomarkers to generate a score that correlates to the degree of liver damage in participants. Scores range from 0 to 1, with higher scores indicating more severe liver fibrosis.
Time Frame: From Day 1 up to 3 years post-treatment
Population: Full Analysis Set (FAS):all participants who received ABT-493 and/or ABT-530 in a prior Phase 2 /3 study and were not retreated prior to enrolling in this study.Three participants who received retreatment prior to enrollment in this study and four participants who did not receive ABT-493 and/or ABT-540 in a prior study were excluded from the FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 367
units on a scale
  Day 1 | 0.354 (0.2341)
  Month 3: number analyzed (Participants) | 347
  Month 3 | 0.363 (0.2383)
  Month 6: number analyzed (Participants) | 333
  Month 6 | 0.353 (0.2311)
  Month 12: number analyzed (Participants) | 2
  Month 12 | 0.405 (0.0919)
  Month 18: number analyzed (Participants) | 5
  Month 18 | 0.272 (0.1281)
  Month 24: number analyzed (Participants) | 227
  Month 24 | 0.321 (0.2156)
  Month 30: number analyzed (Participants) | 68
  Month 30 | 0.261 (0.1667)
  Month 36: number analyzed (Participants) | 1
  Month 36 | 0.190

7. Secondary Outcome: Mean Aspartate Transaminase to Platelet Ratio Index (APRI) Over Time
Description: A serum sample for aspartate transaminase evaluation and platelets were collected at study visits for all participants, until the end of the study or initiation of re-treatment for HCV (if applicable). The aspartate transaminase to platelet ratio index (APRI) is used to assess liver fibrosis in participants with chronic liver disease. Scores range from 0 to ≥ 2.0, with scores < 0.5 predictive of no liver fibrosis; scores >1.5 significant fibrosis; and scores > 2.0 indicative of cirrhosis.
Time Frame: From Day 1 up to 3 years post-treatment
Population: Full Analysis Set (FAS):all participants who received ABT-493 and/or ABT-530 in a prior Phase 2 /3 study and were not retreated prior to enrolling in this study. Three participants who received retreatment prior to enrollment in this study and four participants who did not receive ABT-493 and/or ABT-540 in a prior study were excluded from the FAS.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 367
ratio
  Day 1 | 0.317 (0.2268)
  Month 3: number analyzed (Participants) | 352
  Month 3 | 0.303 (0.2171)
  Month 6: number analyzed (Participants) | 333
  Month 6 | 0.298 (0.2101)
  Month 12: number analyzed (Participants) | 1
  Month 12 | 0.230
  Month 18: number analyzed (Participants) | 5
  Month 18 | 0.262 (0.0589)
  Month 24: number analyzed (Participants) | 232
  Month 24 | 0.275 (0.1620)
  Month 30: number analyzed (Participants) | 69
  Month 30 | 0.227 (0.1084)
  Month 36: number analyzed (Participants) | 2
  Month 36 | 0.215 (0.1768)

8. Secondary Outcome: Mean FibroScan Scores Over Time
Description: The FibroScan test is used to assess liver fibrosis in participants with chronic liver disease. This was not performed as a study procedure, but any available results from source documents were summarized. For participants with Hepatitis C infection, a Fibroscan score of 2-7 kPa indicates no liver scarring or mild scarring; a score of 8 or 9 is associated with moderate liver scarring; 9-14 indicates severe liver scarring; and 14 or higher is indicative of advanced liver scarring, cirrhosis.
Time Frame: Up to 3 years post-treatment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 23
kPa
  Day 1: number analyzed (Participants) | 7
  Day 1 | 13.014 (12.6850)
  Month 3: number analyzed (Participants) | 5
  Month 3 | 6.880 (4.6677)
  Month 6: number analyzed (Participants) | 10
  Month 6 | 10.780 (5.9260)
  Month 12: number analyzed (Participants) | 10
  Month 12 | 7.700 (4.2208)
  Month 18: number analyzed (Participants) | 8
  Month 18 | 6.913 (2.8002)
  Month 24 | 6.757 (3.1564)
  Month 30: number analyzed (Participants) | 1
  Month 30 | 9.400

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) that the investigator considered reasonably related to interventional study procedures or those considered reasonably related to ABT-530 and/or ABT-493 exposure in the prior study by the investigator were collected from the time of the Day 1 visit of the current study period through the last study procedure or discontinuation from study, whichever was later, up to 3 years post-treatment.
Description: An adverse event (AE) in this study is defined as any untoward medical occurrence in a patient or clinical investigation subject that occurs as a result of a study procedure, or is considered by the investigator to be reasonably related to exposure to ABT-493 and/or ABT-530 in the previous study. Deaths were collected as a medical event from the time of informed consent through study end. Serious adverse events outside of the study time frame and all nonserious adverse events were not collected.
Groups:
- HCV-infected Participants-- FAS: Full Analysis Set (FAS): all participants who received ABT-493 and/or ABT-530 in a prior Phase 2 /3 study and were not retreated prior to enrolling in this study. Three participants who received retreatment prior to enrollment in this study and four participants who did not receive ABT-493 and/or ABT-530 in a prior study were excluded from the FAS.
Arm/Group | HCV-infected Participants-- FAS
All-Cause Mortality (participants affected / at risk) | 1/377
Serious Adverse Events (participants affected / at risk) | 0/377
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-10-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT02441283/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT02441283/SAP_001.pdf